CLINICAL TRIAL: NCT00875355
Title: Phase II Randomized Multicenter Study Comparing Brain Radiation in Combination With Temozolomide or Radiation Alone in Patients With Brain Metastases From Breast Cancer
Brief Title: Radiation Therapy With or Without Temozolomide in Treating Women With Brain Metastases and Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institut Curie (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000633496; CLCC-IC-RT-TEMODAL; CLCC-IC-2007-01; INCA-RECF0630; EUDRACT-2007-002531-83; SCHER-CLCC-IC-RT-TEMODAL
Record Dates: First submitted 2009-04-02; First posted 2009-04-03 (Estimated); Last update posted 2009-08-26 (Estimated); Status verified 2009-07

CONDITIONS: Breast Cancer; Metastatic Cancer
Keywords: tumors metastatic to brain; stage IV breast cancer
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis; Brain Neoplasms | interventions — Temozolomide; Radiotherapy

ARMS (2):
- Arm I (Experimental): Patients undergo isocentric radiotherapy to the brain 5 times a week for 2 weeks.
  Interventions: Radiation: radiation therapy
- Arm II (Experimental): Patients undergo radiotherapy as in arm I and receive oral temozolomide once daily for 2 weeks.
  Interventions: Drug: temozolomide; Radiation: radiation therapy

INTERVENTIONS:
Drug: temozolomide — Given orally
  Arms: Arm II
Radiation: radiation therapy — Patients undergo radiotherapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to kill tumor cells. Drugs used in chemotherapy, such as temozolomide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. It is not yet known whether radiation therapy is more effective when given alone or together with temozolomide in treating brain metastases secondary to breast cancer.

PURPOSE: This randomized phase II trial is studying how well radiation therapy given together with temozolomide works compared with radiation therapy given alone in treating women with brain metastases and breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the objective response rate at 6 weeks in women with brain metastases secondary to breast cancer treated with radiotherapy with vs without temozolomide.

Secondary

* Evaluate the tolerability.
* Compare the duration of response.
* Compare local progression-free survival.
* Compare overall survival.

OUTLINE: This is a multicenter study. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients undergo isocentric radiotherapy to the brain 5 times a week for 2 weeks.
* Arm II: Patients undergo radiotherapy as in arm I and receive oral temozolomide once daily for 2 weeks.

After completion of study treatment, patients are followed at 3 and 6 months and then every 6 months for 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of breast cancer

  * Unresectable disease or patient refused surgery
* Must have brain metastases

PATIENT CHARACTERISTICS:

* WHO performance status 0-2
* ANC ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Liver transaminases ≤ 1.5 times upper limit of normal (ULN)
* Creatinine < 1.5 times ULN
* Not pregnant or nursing
* Fertile patients must use effective contraception
* No carcinomatous meningitis
* No history of cancer except for basal cell carcinoma of the skin or carcinoma in situ of the cervix
* No other serious concurrent disease that is, in the opinion of the investigator, likely to interfere with study evaluation and treatment
* No contraindications to treatment with temozolomide
* No psychological, familial, social, or geographic situations that preclude clinical follow up
* No patient deprived of liberty or under guardianship

PRIOR CONCURRENT THERAPY:

* No prior brain radiotherapy
* At least 10 days since prior chemotherapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2007-11; Primary Completion 2009-11 (Estimated)

PRIMARY OUTCOMES:
Response at 6 weeks as assessed by MRI and/or scan

CONTACTS AND LOCATIONS:
Overall Officials: Youlia Kirova, Principal Investigator — Institut Curie
Locations (1):
- Institut Curie Hopital, Paris, France

REFERENCES:
- [Derived] Cao KI, Lebas N, Gerber S, Levy C, Le Scodan R, Bourgier C, Pierga JY, Gobillion A, Savignoni A, Kirova YM. Phase II randomized study of whole-brain radiation therapy with or without concurrent temozolomide for brain metastases from breast cancer. Ann Oncol. 2015 Jan;26(1):89-94. doi: 10.1093/annonc/mdu488. Epub 2014 Oct 29. PMID 25355723